CLINICAL TRIAL: NCT00288106
Title: Prostate Cancer Prevention Trial (PCPT) Companion Long Term Follow Up Study for Men Diagnosed With Prostate Cancer
Brief Title: S0437 Long-Term Follow-Up of Patients Who Were Diagnosed With Prostate Cancer on PCPT
Status: Terminated | Type: Observational
Why Stopped: Poor accrual resulted in lack of feasibility to evaluate endpoints.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000466341; U10CA012027 (NIH); S0437 (Other: SWOG)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Long Term Follow-Up: Follow-up data collection study for men who developed prostate cancer after participation in SWOG-9217 (PCPT)
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — No additional drug was given; clinical observation of men diagnosed with prostate cancer who were previously randomized and treated on PCPT
  Other Names: Observation

SUMMARY:
RATIONALE: Learning about the long-term effects of chemoprevention drugs, such as finasteride, in patients with prostate cancer may help doctors plan better treatment and follow-up care.

PURPOSE: This clinical trial is following patients who were diagnosed with prostate cancer while undergoing treatment with either finasteride or a placebo on the Prostate Cancer Prevention Trial (PCPT).

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to metastases in patients who were diagnosed with high grade or low grade prostate cancer on or before December 31, 2003 and were treated with finasteride or placebo while enrolled on the Prostate Cancer Prevention Trial (SWOG-9217).
* Compare the difference in time to secondary therapy after definitive therapy with radiotherapy or radical prostatectomy in these patients.
* Compare the difference in time to prostate-specific antigen recurrence after definitive therapy with radiotherapy or radical prostatectomy in these patients.
* Compare the difference in all-cause and prostate cancer mortality in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to survival status (alive vs deceased).

Patients provide information about their general health, prostate cancer treatment history, prostate cancer status (i.e., disease progression and metastases data), and prostate-specific antigen (PSA) test results at baseline and then every 6 months for up to 8 years. Next of kin of deceased patients are asked to release the patients' medical records in order to obtain information about the patients' prostate cancer treatment history, prostate cancer progression and metastases, PSA test results, and cause of death.

PROJECTED ACCRUAL: A minimum of 75% of the 2,401 patients (n=1800) diagnosed with prostate cancer on PCPT are needed to have minimal power to evaluate the objectives.

ELIGIBILITY:
INCLUSION CRITERIA:

* Randomized on PCPT
* Diagnosed with prostate cancer on or before December 31, 2003

DISEASE CHARACTERISTICS:

* Diagnosed by either study site or central pathology review

PATIENT CHARACTERISTICS:

* See inclusion criteria

PRIOR CONCURRENT THERAPY:

* Not Applicable

Ages: 55 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men diagnosed with prostate cancer on or before 12/31/03 after participation in the Prostate Cancer Prevention Trial (SWOG-9217)
Sampling Method: Non-Probability Sample
Enrollment: 961 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Time to metastases | Up to 8 years post registration

SECONDARY OUTCOMES:
Time to secondary therapy after definitive therapy | Up to 8 years post registration
  Definitive therapy is defined as radiotherapy or radical prostatectomy.
Time to PSA recurrence after definitive therapy | Up to 8 years post registration
  Definitive therapy is defined as radiotherapy or radical prostatectomy.
All cause and prostate cancer-specific mortality | Up to 8 years post registration
  Measured in a time-to-event analysis

OTHER OUTCOMES:
Predictive value of prognostic biomarkers | Up to 8 years post registration
  To enhance the follow-up for the evaluation of the prognostic biomarkers, which are measured outside the scope of this protocol, on the risk of metastatic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M. Thompson, MD, Study Chair — The University of Texas Health Science Center at San Antonio; Scott M. Lippman, MD, FACP, Study Chair — M.D. Anderson Cancer Center; E. David Crawford, MD, Study Chair — University of Colorado, Denver
Locations (52):
- United States (52):
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Randolph Hospital, Asheboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Danville Regional Medical Center, Danville, Virginia

REFERENCES:
- [Derived] Chau CH, Price DK, Till C, Goodman PJ, Chen X, Leach RJ, Johnson-Pais TL, Hsing AW, Hoque A, Tangen CM, Chu L, Parnes HL, Schenk JM, Reichardt JK, Thompson IM, Figg WD. Finasteride concentrations and prostate cancer risk: results from the Prostate Cancer Prevention Trial. PLoS One. 2015 May 8;10(5):e0126672. doi: 10.1371/journal.pone.0126672. eCollection 2015. PMID 25955319